CLINICAL TRIAL: NCT00000285
Title: Effects of Phenytoin on Cocaine Use in Humans
Brief Title: Effects of Phenytoin on Cocaine Use in Humans - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-2; P50-09259-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Phenytoin

INTERVENTIONS:
Drug: Phenytoin

SUMMARY:
The purpose of this study is to determine the effects of phenytoin on the self-administration of smoked cocaine.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effects of phenytoin on smoked cocaine-base self-administration using our laboratory self-administration model. A total of 12 patients randomized, 6 to phenytoin and 6 to placebo treatment group. There were 2 phases in this 10-day inpatient study. Phase 1 subjects underwent one cocaine self-admin session. Randomization took place at the start of Phase 2, Day 4 where subjects received either placebo or phenytoin. The subjects assigned to phenytoin treatment received an oral loading dose (20mg/kg) aimed at achieving plasma phenytoin concentration of (10-20 mg/L). During Phase 2, subjects had the opportunity to self-administer cocaine on Days 5, 7, and 9. The plasma phenytoin levels were expected to decrease gradually during Phase 2 which provided an opportunity to study the effect of decreasing phenytoin plasma concentrations on cocaine self-administration.

ELIGIBILITY:
Inclusion Criteria:

Males/Females between the ages of 20-40. History of smoked cocaine use on the avg. of at least 2 times/week over a 6 month period. Have currently used at least 1 g of cocaine within a 4-6 hr period. Current history of good health, normal serum albumin levels and normal QTc intervals. Nonreactive for HIV. No participation in any of our studies for the past 6 months. For females: not pregnant as determined by pregnancy screening nor breat feeding, and using acceptable birth control methods (e.g. birth control pills, diaphragm, condoms plus foam).

Exclusion Criteria:

History of suicide attempt, bipolar disorder, schizophrenia, or generalized anxiety disorder. Current problem with major depressive disorder. Current use of alcohol or other durgs on a daily basis. History of major medical illnesses. Currently on parole, probation or a legal history of violence. Treated for chemical dependency within the past 6 months. Use of any psychotropic drugs including MAOIs in the past 6 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-05; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective effects
Physiological effects
Behavioral

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Drug Alcohol Depend. 53:273-75, 1999. Manuscript in preparation.